CLINICAL TRIAL: NCT04324398
Title: Influence of Intra-Canal Cryotherapy on Post-Endodontic Pain and Interleukin-6 Expression Using Different Irrigation Protocols: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Collaborators: Nelly AbdElsalam (Unknown); Dalia Fayyad (Unknown)
Responsible Party: Principal Investigator, Ahmed Emad, principal investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SuezCanalU
Record Dates: First submitted 2020-03-20; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Symptomatic Periapical Periodontitis
Keywords: Cryotherapy; Interleukins; Postoperative pain; Sodium hypochlorite
MeSH Terms: conditions — Pain, Postoperative | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group I (control ) (No Intervention): irrigation with 5% sodium hypochlorite at room temperature from the beginning of cleaning and shaping, between each file and till the final rinse
- Group II (Experimental): irrigation with 5% cold sodium hypochlorite (2-5°C) from the beginning of cleaning and shaping and between each file. Final rinse was done by 20 mL of 5% cold sodium hypochlorite (2-5°C) for 5 minutes
  Interventions: Other: Cryotherapy
- Group III (Experimental): irrigation with 5% sodium hypochlorite at room temperature from the beginning of cleaning and shaping and between each file. Then final rinse with 20 mL of 5% cold sodium hypochlorite (2-5°C) for 5 minutes
  Interventions: Other: Cryotherapy
- Group IV (Experimental): irrigation with 5% sodium hypochlorite at room temperature from the beginning of cleaning and shaping and between each file. Then final rinse with 20 mL of cold saline (2-5°C) for 5 minutes
  Interventions: Other: Cryotherapy

INTERVENTIONS:
Other: Cryotherapy — cold application
  Arms: Group II; Group III; Group IV

SUMMARY:
the study was to evaluate the effect of intra-canal cryotherapy on post-endodontic pain and interleukin-6 expression in teeth with symptomatic apical periodontitis using different irrigation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Anterior or premolar single canal in single rooted teeth.
* Patients aged 20 to 50 years.

Exclusion Criteria:

* Patients under anti-inflammatory medication, immune-suppressive chemotherapy or any antibiotic medication for the last 2 months.
* Pregnant or lactating females.
* Teeth with endo-perio lesions.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
PAIN | one week
  post-operative pain is measured by using visual analogue scale (VAS) The modified VAS will include a 10 cm straight horizontal line numbered at each centimeter with following criteria: (0) for no pain, (1-3) for mild pain, (4-6) for moderate pain, (7-9) for severe tolerable pain and (10) for severe intolerable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed, Port Said, Egypt